CLINICAL TRIAL: NCT02703454
Title: Focal Impulse and Rotor Modulation (FIRM) Ablation Versus Pulmonary Vein Isolation (PVI) for the Treatment of Paroxysmal Atrial Fibrillation (PAF)
Brief Title: FIRM Ablation Versus Pulmonary Vein Isolation for the Treatment of Paroxysmal Atrial Fibrillation (PAF)
Acronym: FIRMAP-AF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLN - 107
Record Dates: First submitted 2016-03-04; First posted 2016-03-09 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FIRM-only (Experimental): Subjects in this arm will be treated with FIRM-guided RF ablation without pulmonary vein isolation (PVI).
  Interventions: Procedure: FIRM-guided RF ablation
- Conventional (Active Comparator): Subjects in this arm will undergo conventional radio frequency (RF) ablation with confirmation of PVI.
  Interventions: Procedure: Conventional RF ablation

INTERVENTIONS:
Procedure: FIRM-guided RF ablation
  Arms: FIRM-only
Procedure: Conventional RF ablation
  Arms: Conventional

SUMMARY:
The study is designed as a prospective, multicenter, single-blind, randomized study to assess the safety and effectiveness of FIRM-guided radiofrequency (RF) ablation procedures for the treatment of symptomatic paroxysmal atrial fibrillation (PAF). The subjects will be blinded to study treatment for the duration of the study period.

ELIGIBILITY:
Key Inclusion Criteria:

* Experiencing at least two (2) documented episodes of paroxysmal atrial fibrillation in the last 3 months preceding study entry with clinical indication for atrial fibrillation (AF) ablation per guidelines. At least one episode should be documented by rhythm strip or ECG.
* Indicated for AF ablation according to current European Heart Rhythm Association (EHRA) guidelines.
* Prescribed with oral anticoagulation therapy, in indicated patients per the latest EHRA guidelines.
* Willingness and able to remain on anti-coagulation therapy as per the latest EHRA guidelines.
* Left atrial diameter < 5.5 cm as measured and image ((computed tomography (CT)/ transesophageal echocardiogram (TEE)/ transthoracic echocardiogram (TTE)/ magnetic resonance imaging (MRI) or intracardiac echocardiography (ICE)) documented within previous six months up to pre-procedure.
* Sustained AF (>5 min uninterrupted) during the electrophysiology procedure. If the subject is not experiencing spontaneous, sustained AF, it may be induced by burst pacing (typically from the coronary sinus) with or without isoproterenol infusion in conventional clinical fashion.

Key Exclusion Criteria:

* New York Heart Association heart failure (NYHA) Class III - IV.
* Ejection fraction < 40% (within previous six months).
* History of myocardial infarction (MI) within the past three months.
* Any concomitant arrhythmia or therapy that could interfere with the interpretation of the results from this study.
* Atrial septal defect (ASD) closure device, left atrial appendage (LAA) closure device, prosthetic mitral or tricuspid valve, or permanent pacemaker.
* Any previous AF catheter ablation.
* History of prior cardioversion for AF lasting > 48 hours.
* Continuous AF episode lasting > 7 days immediately prior to the procedure without a sinus rhythm.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-02; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roland R. Tilz, PD Dr. med., Principal Investigator — Universität zu Lübeck; Phillipp Sommer, PD Dr. med., Principal Investigator — University of Leipzig
Locations (1):
- Universitäres Herzzentrum Lübeck, Lübeck, Germany

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- FIRM-only: Subjects in this arm will be treated with Focal Impulse and Rotor Modulation (FIRM)-guided conventional radio frequency (RF) ablation without pulmonary vein isolation (PVI).
  FIRM-guided RF ablation
- Conventional: Subjects in this arm will undergo conventional RF ablation with confirmation of PVI.
  Conventional RF ablation
Period: Overall Study
Arm/Group | FIRM-only | Conventional
Started | 24 | 27
Treated | 23 | 24
Completed | 13 | 11
Not Completed | 11 | 16
Not completed — Not treated | 1 | 3
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Study discontinuation | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- FIRM-only: Subjects in this arm will be treated with FIRM-guided conventional RF ablation without pulmonary vein isolation (PVI).
  FIRM-guided RF ablation
- Total: Total of all reporting groups
Arm/Group | FIRM-only | Conventional | Total
Number analyzed (Participants) | 24 | 27 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (11.4) | 65 (9.7) | 63 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 14 | 15 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 25 | 49
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 24 | 26 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27 (6.2) | 28 (5.5) | 28 (5.8)
European Heart Rhythm Association (EHRA) symptom classification in atrial fibrillation (AF) [Count of Participants; unit: Participants] — The EHRA score considers symptoms that are attributable to AF and reverse or reduce upon restoration of sinus rhythm or with effective rate control.
  Classification of AF-related symptoms (EHRA score) are as follows:
  EHRA I - 'No symptoms' EHRA II - 'Mild symptoms'; normal daily activity not affected EHRA III - 'Severe symptoms'; normal daily activity affected EHRA IV - 'Disabling symptoms'; normal daily activity discontinued
  Reference:(1) Eur Heart J. 2010 (19):2369-429
  Participants
    Class I | 2 | 0 | 2
    Class II | 8 | 7 | 15
    Class III | 14 | 18 | 32
    Class IV | 0 | 1 | 1
    Unknown | 0 | 1 | 1
History of Arterial Hypertension [Count of Participants; unit: Participants]
  Yes | 11 | 13 | 24
  No | 9 | 8 | 17
  Unknown | 4 | 6 | 10
History of Coronary Artery Disease [Count of Participants; unit: Participants]
  Yes | 8 | 8 | 16
  No | 12 | 13 | 25
  Unknown | 4 | 6 | 10
History of Chronic Renal Insufficiency [Count of Participants; unit: Participants]
  Yes | 2 | 3 | 5
  No | 18 | 18 | 36
  Unknown | 4 | 6 | 10
Left Atrial Diameter [Mean (Standard Deviation); unit: mm] | 44 (5.5) | 44 (7.3) | 44 (6.4)
Anti-Arrhythmic Use at Baseline: Amiodarone [Count of Participants; unit: Participants]
  Yes | 2 | 0 | 2
  No | 22 | 25 | 47
  Unknown | 0 | 2 | 2
Anti-Arrhythmic Use at Baseline: Dronedarone [Count of Participants; unit: Participants]
  Yes | 0 | 0 | 0
  No | 24 | 25 | 49
  Unknown | 0 | 2 | 2
Anti-Arrhythmic Use at Baseline: Flecainide [Count of Participants; unit: Participants]
  Yes | 4 | 7 | 11
  No | 20 | 18 | 38
  Unknown | 0 | 2 | 2
Anti-Arrhythmic Use at Baseline: Propafenone [Count of Participants; unit: Participants]
  Yes | 1 | 0 | 1
  No | 23 | 25 | 48
  Unknown | 0 | 2 | 2
Anti-Arrhythmic Use at Baseline: Sotalol [Count of Participants; unit: Participants]
  Yes | 0 | 2 | 2
  No | 24 | 23 | 47
  Unknown | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Single-procedure Freedom From AF/AT Recurrence From 3-12 Months Post Index Ablation Procedure
Description: Freedom from AF/AT recurrence is defined as no documented episodes of AF/AT > 30 seconds with conventional non-invasive monitoring. In the case of a cardiac implanted electronic device (CIED), freedom from AF recurrence is defined as no documented episodes of AF/AT > 30 seconds in a 72-hour window at the follow-up visits in addition to any symptomatic episodes with documented AF > 30 seconds. AT recurrence does not include episodes of cavotricuspid isthmus (CTI) dependent flutter.
Time Frame: 3 -12 months post study treatment.
Population: Patients with 12-month follow-up data
Measure: Count of Participants; unit: Participants
Arm/Group | FIRM-only | Conventional
Number analyzed (Participants) | 16 | 10
Participants | 5 | 8

2. Secondary Outcome: Number of Participants With Freedom From Procedure-related Serious Adverse Events
Description: Freedom from procedure-related serious adverse events within one year of the index procedure
Time Frame: Within 1 year post study treatment
Population: Subjects with 12 month safety data
Measure: Count of Participants; unit: Participants
Arm/Group | FIRM-only | Conventional
Number analyzed (Participants) | 15 | 14
Participants | 12 | 14

ADVERSE EVENTS:
Time Frame: Adverse event data was collected up to 1 year post index procedure.
Arm/Group | FIRM-only | Conventional
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/27
Serious Adverse Events (participants affected / at risk) | 12/24 | 4/27
Other Adverse Events (participants affected / at risk) | 4/24 | 1/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FIRM-only (N=24) | Conventional (N=27)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0)
Accidental Exposure to Product (General disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Aneurysma Aorta Ascendens (Vascular disorders) | 0 (0) | 1 (1)
Aortic Valve Stenosis (Vascular disorders) | 0 (0) | 1 (1)
Atrial Tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
Bleeding Aneamia (Vascular disorders) | 0 (0) | 1 (1)
Blood Sodium Decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Carotid Artery Stenosis (Vascular disorders) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 1 (1)
Cerebral Infarction (Vascular disorders) | 0 (0) | 1 (1)
Chondromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Coronary Artery Disease (Vascular disorders) | 0 (0) | 1 (1)
Femoral Artery Occlusion (Vascular disorders) | 0 (0) | 1 (1)
Femoral Artery Aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Fracture Of Distale Radius Left, Orbita And Maxillary Sinus (General disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Haematoma, Injection Site (Vascular disorders) | 2 (2) | 0 (0)
Haematoma, Right Groin (Vascular disorders) | 1 (1) | 0 (0)
Liver Abscess (Hepatobiliary disorders) | 1 (1) | 0 (0)
Phrenic Nerve Paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Occlusion Of Arteria Femoralis Pop-Iii-Bypass Right Side (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Syncope (Vascular disorders) | 0 (0) | 2 (2)
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Suspected Dementia With Hospitalisation Due To Diagnostic Tests (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FIRM-only (N=24) | Conventional (N=27)
Atrial Fibrillation (Cardiac disorders) | 4 (4) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination led to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The data and results from this study are the sole property of Sponsor. Investigators will not use data from this clinical investigation without the written consent of the Sponsor or generate publication materials as referenced in the Clinical Trial Agreement Single-center results are not allowed to be published or presented before the multi-center results.

DOCUMENTS (2):
  • Study Protocol (2015-12-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT02703454/Prot_000.pdf
  • Statistical Analysis Plan (2016-01-05): https://cdn.clinicaltrials.gov/large-docs/54/NCT02703454/SAP_001.pdf